CLINICAL TRIAL: NCT00551863
Title: Development of Violence Therapy for Substance Abusers
Brief Title: Developing Violence Prevention Therapy for Substance Abusers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Chermack, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA017295-01A1 (NIH); R01DA017295 (NIH)
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Substance Use Disorders; Violence
Keywords: alcohol, drugs, aggression, substance use disorder treatment
MeSH Terms: conditions — Substance-Related Disorders; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVPT (Active Comparator): Intervention based on Motivational Interviewing and CBT
  Interventions: Behavioral: IVPT

INTERVENTIONS:
Behavioral: IVPT — Violence prevention intervention based on Motivational Interviewing and CBT

SUMMARY:
The purpose of this project is to develop and pilot test a violence prevention intervention for men and women in treatment for substance use problems.

ELIGIBILITY:
Inclusion Criteria:

* Presence of substance use related problems
* Interpersonal Violence history in the year before recruitment

Exclusion Criteria:

* Primary opiate dependence
* Presence of active psychotic disorder
* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Interpersonal Violence | 3 and 6 month follow-up

SECONDARY OUTCOMES:
alcohol and drug use | 3 and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Chermack, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Epstein-Ngo QM, Walton MA, Sanborn M, Kraus S, Blow F, Cunningham R, Chermack ST. Distal and proximal factors associated with aggression towards partners and non-partners among patients in substance abuse treatment. J Subst Abuse Treat. 2014 Oct;47(4):282-92. doi: 10.1016/j.jsat.2014.05.005. Epub 2014 Jun 10. PMID 25012548
- [Background] Ilgen MA, Chermack ST, Murray R, Walton MA, Barry KL, Wojnar M, Blow FC. The association between partner and non-partner aggression and suicidal ideation in patients seeking substance use disorder treatment. Addict Behav. 2009 Feb;34(2):180-6. doi: 10.1016/j.addbeh.2008.10.004. Epub 2008 Oct 10. PMID 18977093
- [Background] Chermack ST, Murray RL, Winters JJ, Walton MA, Booth BM, Blow FC. Treatment needs of men and women with violence problems in substance use disorder treatment. Subst Use Misuse. 2009;44(9-10):1236-62. doi: 10.1080/10826080902960007. PMID 19938916
- [Background] Murray RL, Chermack ST, Walton MA, Winters J, Booth BM, Blow FC. Psychological aggression, physical aggression, and injury in nonpartner relationships among men and women in treatment for substance-use disorders. J Stud Alcohol Drugs. 2008 Nov;69(6):896-905. doi: 10.15288/jsad.2008.69.896. PMID 18925348
- [Background] Chermack ST, Murray RL, Walton MA, Booth BA, Wryobeck J, Blow FC. Partner aggression among men and women in substance use disorder treatment: correlates of psychological and physical aggression and injury. Drug Alcohol Depend. 2008 Nov 1;98(1-2):35-44. doi: 10.1016/j.drugalcdep.2008.04.010. Epub 2008 Jun 13. PMID 18554825
- [Background] Chermack ST, Grogan-Kaylor A, Perron BE, Murray RL, De Chavez P, Walton MA. Violence among men and women in substance use disorder treatment: a multi-level event-based analysis. Drug Alcohol Depend. 2010 Dec 1;112(3):194-200. doi: 10.1016/j.drugalcdep.2010.06.005. Epub 2010 Jul 27. PMID 20667666
- [Result] Chermack ST, Bonar EE, Ilgen MA, Walton MA, Cunningham RM, Booth BM, Blow FC. Developing an Integrated Violence Prevention for Men and Women in Treatment for Substance Use Disorders. J Interpers Violence. 2017 Feb;32(4):581-603. doi: 10.1177/0886260515586369. Epub 2016 Jul 11. PMID 26002873